CLINICAL TRIAL: NCT02457195
Title: Preoperative Use of Granisetron Transdermal Patch for Prevention of Postoperative Nausea and Vomiting (PONV) in Patients With History of Severe PONV - Open Label, Prospective, Pilot Study
Brief Title: Granisetron Transdermal Patch for Prevention of Postoperative Nausea and Vomiting
Acronym: GTPPONV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Piotr K Janicki MD, PhD, Professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRP-592
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; anesthesia; granisetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Admnistration of granisetron (Experimental): Preoperative administration of granisetron transdemal patch
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — Application granisetron transdermal patch preoperatively
  Other Names: Sancuso

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of adding transdermal preparation of granisetron (Sancuso ®) to the current postoperative nausea and vomiting (PONV) standard prophylaxis regimen with dexamethasone and ondansetron in patients with the previous history of severe, particularly delayed and/or post-discharge, PONV and undergoing surgical procedure under general anesthesia.

The specific aims of the study include:

1. efficacy of the investigated therapy in prevention of PONV up to 120 hours after surgery
2. incidence and seriousness of the observed side effects
3. ability of patients to self-administer preoperatively and maintain the investigated patch during the perioperative period
4. level of satisfaction with the preoperative PONV prophylaxis.

DETAILED DESCRIPTION:
Patients will be recruited from the surgical population undergoing preoperative evaluation in Anesthesiology Preoperative Evaluation Clinic at Hershey Med. Ctr. (~15,000 per year). Selected patients (ASA 1-3, N=60) with history of severe PONV after one or more of previous general anesthesia, and scheduled to undergo surgical procedures with general anesthesia will be enrolled into IRB approved protocol. The patch will be placed by the patient at home 24 - 48 hours before surgery as directed by the doctor. The subsequent standardized general anesthesia protocol for elective surgery will include general endotracheal anesthesia with sevofluran, including standard intraoperative PONV prophylaxis (IV dexamethasone and IV ondansetron, each 4 mg). Postoperative evaluation will include recording of incidence and severity of PONV at the time of discharge from PACU (acute PONV), at 24 hr, 48 hrs, 72 and 120 hrs (delayed or post discharge PONV).

7.2.1 Visit 1 - Anesthesia Preoperative Evaluation Clinic and recruitment and drug dispensation Patient is seen in clinic and identified as having a history of serious PONV, in particular delayed or post discharge PONV. Study will be explained to the patient and consent obtained. The investigational pharmacy will be notified that a study patient has been enrolled and they will prepare the patches for distribution to the patient.

A member of the research team will obtain the assigned patches from the investigational pharmacy and deliver to the anesthesia provider (member of the research team).

The provider will then demonstrate to the patient how to apply the patch and the patient can practice using a placebo patch to show that the correct placement. Patient will then take the actual patch home with them.

7.2.2 Visit 2 - approximately 24-48 hours preoperatively (patient's home) Patient will apply the patch to their upper arm 24-48 hours before scheduled surgical procedure, as instructed during their pre-op anesthesia visit. The patch will then remain in place until 120 hours after surgical procedure. No backup patch will be provided so the patients with the accidently missing patch will need to call their primary surgical service for the standard antiemetic medication.

7.2.3 Visit 3- Day of Surgery Patient will arrive for surgery. A member of the research team will meet them in the SDU and record the time that the patch was applied, and if it has been placed correctly, intact and still in place. Any potential side effects (systemic or local) will be recorded at that time. The subsequent standardized general anesthesia protocol for elective surgery will include general endotracheal anesthesia with sevofluran (no nitrous oxide), muscle relaxants (with reversal), intraoperative IV opioid analgesics, including standard PONV prophylaxis (dexamethasone and ondansetron IV 4 mg).

Early postoperative evaluation will include recording of incidence and severity of PONV at the time of discharge from PACU (acute PONV). The incidence of vomiting or retching will recorded by the nursing staff. Patients with symptoms requiring a rescue antiemetic-nausea score ≥4 on an 11-point Numeric Rating Scale (NRS), retching or vomiting, or patient request-within 6 hours of PACU admission will be given the rescue medication (Benadryl or promethazine). The NRS was an 11-point linear scale on which patients rated their nausea, with 0 meaning no nausea and 10 meaning the worst possible nausea.

The subsequent evaluations will be performed either at the patient's bed (if in the hospital) or by phone call at 24 hr, 48 hrs, 72 and 120 hrs (delayed or post discharge PONV). The patient will be supplied with a diary to record the information that will be requested on the follow-up phone calls.

The primary efficacy endpoint will be complete response (CR), defined as no emetic episode and no rescue medication; the proportions of patients with no emesis and no additional rescue medication in the 120 hours following the completion of surgical procedure and the change from baseline nausea score using the NRS. Treatment-emergent adverse events (TEAEs), regardless of suspected causal relationship to the study medication, will be also recorded throughout and continued until 5 days after surgery.

7.3 Duration of Participation Patient will remain in the study until all time points have been met (maximum 5 days following surgery or 120 hours). At the end of the study the patient will remove and dispose the remaining patch.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are between the ages of 18 and 89
* Scheduled to undergo surgical procedures with general anesthesia
* Seen in the anesthesia clinic at least 24 hours before surgery
* History of severe PONV after previous general anesthesia
* Surgical procedures with anticipated duration > 1 hour and no more than 5 hours
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Allergy to granisetron or other 5HT3RA drugs
* Previous allergic reactions to any drug skin patches
* Recent (less than 1 month) or current chemo- or radiotherapy
* Any nausea, vomiting, or retching within 24 hours prior to anesthesia
* Any type of eye surgeries
* History or diagnosis of gastrointestinal obstruction or ileus
* History of serotonin syndrome
* Unable to sign consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr K Janicki, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Admnistration of Granisetron
Started | 50
Completed | 41
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Admnistration of Granisetron
Number analyzed (Participants) | 50
Age, Customized [Number; unit: participants]
  18-21 years : female | 0
  18-21 years : male | 0
  22-29 years : female | 2
  22-29 years : male | 0
  30-39 years : female | 5
  30-39 years : male | 0
  40-49 years : female | 13
  40-49 years : male | 0
  50-59 years : female | 11
  50-59 years : male | 2
  60-69 years : female | 13
  60-69 years : male | 0
  70-79 years : female | 3
  70-79 years : male | 0
  80-89 years : female | 1
  80-89 years : male | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 1
  Unknown or Not Reported | 1
Baseline Participants who completed study [Count of Participants; unit: Participants]
  18-21 years : female | 0
  18-21 years : male | 0
  22-29 years : female | 2
  22-29 years : male | 0
  30-39 years : female | 5
  30-39 years : male | 0
  40-49 years : female | 13
  40-49 years : male | 0
  50-59 years : female | 5
  50-59 years : male | 2
  60-69 years : female | 11
  60-69 years : male | 0
  70-79 years : female | 2
  70-79 years : male | 0
  80-89 years : female | 1
  80-89 years : male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR), No PONV Symptoms, Nausea
Description: Composite measure consisting of complete response (CR), defined as no emetic episode and no rescue medication; the proportions of patients with no emesis and no additional rescue medication in the 120 hours following the completion of surgical procedure.
Time Frame: 24 hrs, 48 hrs, 72 hrs and 120 hrs
Population: Those that completed the current study
Measure: Count of Participants; unit: Participants
Groups:
- Admnistration of Granisetron: Outcomes measured in the study patients after application of transdermal granisetron patch throughout the study period
Arm/Group | Admnistration of Granisetron
Number analyzed (Participants) | 41
Participants
  Completed Response : 24 hrs | 8
  Completed Response : 48 hrs | 25
  Completed Response : 72 hrs | 24
  Completed Response : 120 hrs | 28
  No PONV symptoms : 24 hrs | 18
  No PONV symptoms : 48 hrs | 25
  No PONV symptoms : 72 hrs | 24
  No PONV symptoms : 120 hrs | 28
  Nausea : 24 hrs | 21
  Nausea : 48 hrs | 11
  Nausea : 72 hrs | 7
  Nausea : 120 hrs | 3
  Vomiting with or without retching : 24 hrs | 5
  Vomiting with or without retching : 48 hrs | 2
  Vomiting with or without retching : 72 hrs | 0
  Vomiting with or without retching : 120 hrs | 0
  Retching (dry-hives, without vomiting) : 24 hrs | 3
  Retching (dry-hives, without vomiting) : 48 hrs | 1
  Retching (dry-hives, without vomiting) : 72 hrs | 0
  Retching (dry-hives, without vomiting) : 120 hrs | 0

ADVERSE EVENTS:
Time Frame: 120 hours
Description: Granisetron transdermal patch is already FDA approved for treatment of patients with cancer during chemotherapy but has not been tested for treating PONV caused by general anesthesia.
Arm/Group | Admnistration of Granisetron
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 13/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Admnistration of Granisetron (N=50)
skin irritation (Skin and subcutaneous tissue disorders) | 6 — Skin irritation
constipation (Gastrointestinal disorders) | 2 — constipation
diarrhea (Gastrointestinal disorders) | 1 — Diarrhea
hallucination (Nervous system disorders) | 1 — Hallucination
dizziness (General disorders) | 1 — Dizziness
headache (General disorders) | 1 — Headache
EKG changes (Cardiac disorders) | 1 — EKG changes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT02457195/Prot_SAP_000.pdf